CLINICAL TRIAL: NCT05499429
Title: Clinical Single-center Randomized Controlled Trial of Non-invasive Transcranial Focused Low-intensity Ultrasound Stimulation in Patients With Mild Lewy Body Dementia
Brief Title: Non-invasive Transcranial Focused Low-intensity Ultrasound Stimulation in Patients With Mild Lewy Body Dementia
Acronym: tFUS in DLB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2022]110
Record Dates: First submitted 2022-07-14; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Lewy Body Dementia
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to the active stimulation group and sham stimulation group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients were randomly assigned to the active stimulation group and sham stimulation group, Patients，Care Provider and Outcomes Assessor did not know the patient grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stimulus group (Active Comparator): Patients were assigned into active stimulus group according to random number table
  Interventions: Device: Transcranial low intensity focused ultrasound stimulation
- sham stimulus control group (Sham Comparator): Patients were assigned into sham stimulus control group according to random number table
  Interventions: Device: Transcranial low intensity focused ultrasound stimulation

INTERVENTIONS:
Device: Transcranial low intensity focused ultrasound stimulation — Low intensity focused transcranial ultrasound stimulation can safely and effectively regulate neuron excitability through mechanical force.
  Other Names: tFUS

SUMMARY:
A randomized controlled clinical study was conducted in the xuanwu hospital Single Center of Capital Medical University to preliminarily explore the efficacy and safety of transcranial focused low-intensity ultrasound stimulation in the treatment of dementia with Lewy bodies in the early stage, to clarify the effective mechanism and form an effective clinical treatment plan.

DETAILED DESCRIPTION:
This project plans to recruit 20 patients with mild Lewy body dementia.They were randomly divided into transcranial focused low-intensity ultrasound active stimulation group and sham stimulation group. Patients receive treatment three days a week, and the daily treatment time is 20-30 minutes.The duration of treatment is 4-12 weeks. Before treatment, cognitive assessment, resting EEG, head MRI and PET examination of glucose metabolism were completed.Complete the overall cognitive assessment, resting EEG and MRI examination within one week after the treatment, and complete the overall cognitive assessment and PET examination of glucose metabolism at the follow-up 6 months after the treatment.Fill in the treatment side effect scale and adverse event form.Keep the original oral drug dosage unchanged during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Male or female DLB patients between the ages of 50-85;
* The psychological evaluation was in accordance with MMSE score of 18-24 (including 18 and 24) and CDR score of 0.5.
* Can cooperate to complete clinical research.

Exclusion Criteria:

* There is a definite history of cerebrovascular stroke, and there are definite symptoms or signs of neurological deficit at the time of onset, and there are corresponding responsible lesions left by neuroimaging。
* Those who have a history of alcoholism, or drug addiction, or neurological diseases such as brain trauma, epilepsy, encephalitis, normal intracranial pressure hydrocephalus, etc. that can cause cognitive impairment.
* Suffering from systemic diseases that may lead to cognitive impairment (such as liver and kidney insufficiency, endocrine diseases, vitamin deficiency).
* Have a history of using antipsychotics for more than five years before diagnosis.
* There are contraindications for head MRI examination.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale | 12 weeks
  Evaluate the improvement of clinical symptoms.

SECONDARY OUTCOMES:
resting EEG | 12 weeks
  EEG power in alpha band
head MRI | 12 weeks
  Changes of brain function by fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

IPD SHARING:
Plan to Share IPD: No